CLINICAL TRIAL: NCT02146651
Title: A Double-blinded, Randomised, Four-period Crossover Euglycemic Clamp Trial Investigating the Dose-response and Dose-exposure Relationship of BioChaperone Insulin Lispro in Three Different Doses in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BC3-CT008
Record Dates: First submitted 2014-05-20; First posted 2014-05-26 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BioChaperone insulin lispro 0.2U/Kg (Experimental): BioChaperone insulin lispro 0.2U/Kg
  Interventions: Drug: BioChaperone insulin lispro 0.2U/Kg; Drug: BioChaperone insulin lispro 0.1U/Kg; Drug: BioChaperone insulin lispro 0.4U/Kg; Drug: Humalog®
- BioChaperone insulin lispro 0.1U/Kg (Experimental): BioChaperone insulin lispro 0.1U/Kg
  Interventions: Drug: BioChaperone insulin lispro 0.2U/Kg; Drug: BioChaperone insulin lispro 0.1U/Kg; Drug: BioChaperone insulin lispro 0.4U/Kg; Drug: Humalog®
- BioChaperone insulin lispro 0.4U/Kg (Experimental): BioChaperone insulin lispro 0.4U/Kg
  Interventions: Drug: BioChaperone insulin lispro 0.2U/Kg; Drug: BioChaperone insulin lispro 0.1U/Kg; Drug: BioChaperone insulin lispro 0.4U/Kg; Drug: Humalog®
- Humalog® 0.2U/Kg (Active Comparator): Humalog® 0.2U/Kg
  Interventions: Drug: BioChaperone insulin lispro 0.2U/Kg; Drug: BioChaperone insulin lispro 0.1U/Kg; Drug: BioChaperone insulin lispro 0.4U/Kg; Drug: Humalog®

INTERVENTIONS:
Drug: BioChaperone insulin lispro 0.2U/Kg — Single dose of 0.2U/Kg body weight injected subcutaneously
Drug: BioChaperone insulin lispro 0.1U/Kg — Single dose of 0.1U/Kg body weight injected subcutaneously
Drug: BioChaperone insulin lispro 0.4U/Kg — Single dose of 0.4U/Kg body weight injected subcutaneously
Drug: Humalog® — Single dose of 0.2U/Kg body weight injected subcutaneously

SUMMARY:
The addition of BioChaperone to insulin lispro may accelerate the onset and shorten the duration of action of insulin lispro due to facilitation of the absorption of the insulin after subcutaneous injection.

The aim of the trial is to investigate the dose-response and the dose-exposure relationships of BioChaperone insulin lispro under 3 doses, to compare the pharmacokinetics and glucodynamic action of BioChaperone insulin lispro at 0.2U/Kg with Humalog® at 0.2 U/Kg and to assess safety and tolerability of BioChaperone insulin lispro and Humalog®.

This is a double-blinded, randomised, four-period crossover phase 2 trial using automated 12-hour euglycemic clamps in subject with type 1 diabetes mellitus.

Each subject will be randomly allocated to a sequence of 4 treatments, i.e. with one of three single doses of BioChaperone insulin lispro (0.1, 0.2 and 0.4 U/Kg) or one single dose of Humalog® (0.2 U/Kg) on 4 separate dosing visits.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus for at least 12 months
* Treated with multiple daily insulin injections of insulin pump for at least 12 months
* Body Mass Index (BMI): 18.5-28.0 Kg.m²

Exclusion Criteria:

* Type 2 diabetes mellitus
* Receipt of any investigational product within 3 months prior first dosing
* Clinically significant abnormalities as judged by the investigator
* Any systemic treatment with drugs known to interfere with glucose metabolism
* History of alcoholism or drug/chemical abuse as per investigator's judgement
* Use of tobacco or nicotine-contained product within 1 year prior to screening
* Blood or plasma donation in the past month or more than 500ml within 3 months prior to screening

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-05; Primary Completion 2014-07 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Glucodynamic endpoint: Area Under the Curve GIR(0-last) | 12 hours
  Area under the Glucose Infusion Rate time curve from 0 hours until the end of the clamp
Glucodynamic endpoint: GIRMax | 12 hours
  Maximum Glucose Infusion Rate
Pharmacokinetic endpoint: AUC Lisp(0-last) | 12 hours
  Area under the insulin lispro serum concentration - time curve over the clamp procedure.
Pharmacokinetic endpoint: Cmax(Lisp) | 12 hours
  Maximum observed serum insulin lispro concentration

SECONDARY OUTCOMES:
Pharmacokinetics: Tmax(lisp) | 12 hours
  Time to maximum observed serum insulin lispro concentration
Glucodynamic: TGIRmax | 12 hours
  Time to maximum Glucose Infusion Rate
Tonset of action | 12 hours
  Time from t=0 until blood glucose concentration has decreased by 5mg.dL (0.3mmol.L) from baseline.
Safety and Tolerability: adverse events, local tolerability, vital signs variations, ECG, laboratory safety parameters. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil Institut für Stoffwechselfforschung GmbH
Locations (1):
- Profil Institut für stoffwechselforschung GmbH, Neuss, Germany